CLINICAL TRIAL: NCT02417545
Title: Gaze and Movement Behavior of Patients With Vestibular Dysfunction During Level Floor, Ramp, and Stair Walking
Brief Title: Gaze and Stair Walking in Patients With Vestibular Dysfunction
Acronym: Gaze
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-2014-0509
Record Dates: First submitted 2015-04-10; First posted 2015-04-15 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Vestibular Diseases
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to assess the differences in gaze and gait during the stair and ramp negotiation (+transition to normal level walking) between healthy controls and vestibular patients (fallers and non-fallers).

DETAILED DESCRIPTION:
For a better understanding of falls in patients with vestibular disorders it might be important to identify the challenging environmental that provoke functional deficits; e.g. stair or ramp negotiation. The three steps at the ground and at the top of stairs is the most common location for missteps and stair accidents. This is supported by the observation made in a 12-month prospective study were 32% of the falls happened during the last step going down stairs in vestibular patients.

It remains open if patient's vestibular dysfunctions have a different gaze or gait behavior than healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* All included patients are diagnosed with single or two-sided vestibular dysfunction.
* Adult male and female participant's (≥18 years)
* Signed informed consent after being informed

Exclusion Criteria:

* Benign paroxysmal positional vertigo
* Acute pain
* Walking disability (independent walking distance <10 meters)
* Uncontrolled cardiovascular disease (e.g.: uncontrolled blood pressure)
* Gait problems caused by Hip or knee endoprothesis
* Weakness due to neurological problems
* Known or suspected non-compliance
* Contraindications on ethical grounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study sample includs patients with vestibular disorder and age matched healthy participants. Patients with vestibular disorder will be diagnosed by a pathological horizontal head impulse test to both sides (< 0.80), as assessed by using a video-based system and the presents of saccades.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Gaze | 30 minutes
  A mobile eye tracker (Dikablis Professional Glasses, Ergoneers Inc., Manching, Germany) was used to record gaze during the stairs and ramp negotiation.

SECONDARY OUTCOMES:
Gait | 30 minutes
  The recording gait system is a pair of inlay soles with sensors. The sensors sampled the force distribution beneath the subjects' feet. The inlay soles are recording acceleration, rotation rates and magnetic field readings, each in 3 dimensions.
Fall Calendar | one year
  A fall-Calendar with questions will be used to assess falls. These questions will be placed on each page of a 12 month calendar. The "fall calendar" pages also contain questions about the circumstances surrounding falls, including the day time, lighting situation, fall location, activity performed, injuries and whether medical assistance was needed. As soon as possible after the fall the fallers have to fill in the date of the fall, its cause, and fall-related injuries. At the end of each month, a calendar page should be sent by each patient to the investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Swanenburg, PhD, Principal Investigator — University Hospital Zurich, Directorate of Research and Education, Physiotherapy & Occupational Therapy Research
Locations (1):
- University Hospital Zurich, Directorate of Research and Education, Physiotherapy & Occupational Therapy Research, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Publication